CLINICAL TRIAL: NCT03888456
Title: Effects of Osteopathic Manipulative Treatment on Autonomic Nervous System: a Thermography Study
Brief Title: Effects of OMT on ANS: a Thermography Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Come Collaboration (Other)
Collaborators: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other); Chinesis IFOP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: COME-02-18
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Autonomic Nervous System Imbalance; Healthy
MeSH Terms: interventions — Manipulation, Osteopathic; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: randomised placebo controlled crossover study
Who Masked: Participant, Outcomes Assessor
Masking Description: participants will be blindly assigned to study or control arm using a computer-based random sequence generation and seal envelop
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Experimental): participants will receive a single touch intervention based on osteopathic assessment and treatment
  Interventions: Other: osteopathic treatment; Other: sham
- Control (Sham Comparator): participants will receive a single touch sham intervention mimicking the intervention
  Interventions: Other: osteopathic treatment; Other: sham

INTERVENTIONS:
Other: osteopathic treatment — the intervention will be based on 2 phases: 1) assessment to identify areas with somatic dysfunction, 2) treatment to improve the function of the area identified
Other: sham — the sham intervention will consists of 2 overlapping phases as the intervention group but without applying any technique

SUMMARY:
the study will investigate the effect of a specific type of touch intervention on the activity of autonomic nervous system measured using thermography

ELIGIBILITY:
Inclusion Criteria:

* adults above 18y and below 35y
* without any congenital, genetical and chronic disease
* without any symptomatology

Exclusion Criteria:

* congenital, genetical and chronic disease
* neurological, cardiovascular, psychiatric disease
* acute pain
* paediatric patients
* adults over 35 years old

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
temperature | 1 week
  variability of the autonomic nervous system measured by temperature variability of the face

SECONDARY OUTCOMES:
skin conductance | 1 week
  pre-post changes of physiological parameter of electrodermal skin response
heart rate variability | 1 week
  pre-post changes of HRV

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cerritelli, Principal Investigator — Come Collaboration
Locations (1):
- University of Chieti, Chieti, Italy

REFERENCES:
- [Derived] Cerritelli F, Cardone D, Pirino A, Merla A, Scoppa F. Does Osteopathic Manipulative Treatment Induce Autonomic Changes in Healthy Participants? A Thermal Imaging Study. Front Neurosci. 2020 Aug 18;14:887. doi: 10.3389/fnins.2020.00887. eCollection 2020. PMID 33013294